CLINICAL TRIAL: NCT01245504
Title: Clinical Evaluation of an Algorithm to Assess Sockets Made by Central Fabrication Facilities
Brief Title: Assessment of Socket Shapes Made by Central Fabrication Facilities
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Joan Sanders, Professor, University of Washington
Other Study IDs: 31673 E/B
Record Dates: First submitted 2010-11-18; First posted 2010-11-22 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: People With Lower Limb Amputation That Are Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lower-limb amputee: Subjects with at least one lower limb amputated at teh trans-tibial level
  Interventions: Other: Assessed for socket fit

INTERVENTIONS:
Other: Assessed for socket fit — Subjects are clinically assessed during standing to see how well computer manufactured sockets fit

SUMMARY:
Quality and accuracy of prosthetic sockets manufactured by central fabrication facilities may be lacking. Poor quality manufacturing can be detrimental to socket fit in amputees and may require more work by prosthetists to redesign the socket. The aim of this research is to assess the accuracy of prosthetic sockets manufactured by commercial companies. Determination of how and where manufacturing errors occur will contribute to better quality of socket fit for the amputee patient and improve the efficiency of prosthetists who fit the manufactured products to their patients.

Computer manufactured sockets are made for subjects, then their fits assessed by research practitioners.

ELIGIBILITY:
Inclusion Criteria:

* trans-tibial amputees who use a prosthesis and are ambulatory

Exclusion Criteria:

* do not have a prosthesis, cannot ambulate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: people with lower limb amputation that are ambulatory
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Limb volume | 1 day

SECONDARY OUTCOMES:
Limb shape | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Bioengineering Department, Seattle, Washington, United States